CLINICAL TRIAL: NCT01550276
Title: Treatment of Tension-type Headache With Articulatory and Suboccipital Soft Tissue Therapy: a Double-blind, Randomized, Placebo-controlled Clinical Trial
Brief Title: Treatment of Tension-type Headache With Articulatory and Suboccipital Soft Tissue Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, GEMMA V ESPÍ LÓPEZ, PhD, PhD, PT, University of Valencia
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: UVT001
Record Dates: First submitted 2012-02-15; First posted 2012-03-09 (Estimated); Last update posted 2012-03-09 (Estimated); Status verified 2012-03

CONDITIONS: Tension-type Headache
Keywords: Effectiveness; Tension-type headache; Manual therapy
MeSH Terms: conditions — Tension-Type Headache | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Suboccipital soft tissue inhibition (Experimental): The SI treatment aims to release the suboccipital muscle spasm that maintains the occiput-atlas-axis joint dysfunction.
  Interventions: Other: Manual Therapy
- Occiput-atlas-axis global manipulation (Experimental): The OAA manipulation was bilaterally administered and it attempts to restore the motion dysfunction of this complex
  Interventions: Other: Manual Therapy
- The combination of both treatments (Experimental)
  Interventions: Other: Manual Therapy
- control group (Placebo Comparator)
  Interventions: Other: Placebo control

INTERVENTIONS:
Other: Manual Therapy — All patients were assessed in the same conditions before the treatment, after the treatment (at 4 weeks), and at follow-up (after 8 weeks). Four treatment sessions (one session per week). Prior to each treatment session, the physiotherapist performed the vertebral artery test bilaterally, followed by a two-minute neck massage without lubricants and with no proven therapeutic effect, as a placebo for all study groups.
  The SI treatment aims to release the suboccipital muscle spasm10 that maintains the occiput-atlas-axis joint dysfunction. This technique, which was administered for 10 minutes, uses a deep and progressive gliding pressure applied with the fingertips towards the posterior arch of atlas.
  Arms: Suboccipital soft tissue inhibition
Other: Manual Therapy — All patients were assessed in the same conditions before the treatment, after the treatment (at 4 weeks), and at follow-up (after 8 weeks). Four treatment sessions (one session per week). Prior to each treatment session, the physiotherapist performed the vertebral artery test bilaterally, followed by a two-minute neck massage without lubricants and with no proven therapeutic effect, as a placebo for all study groups.
  The OAA manipulation was bilaterally administered and it attempts to restore the motion dysfunction of this complex. It is a structural technique performed on a vertical line along the odontoid process of axis; neither flexion nor extension is used, and lateroflexion is minimal.
  Arms: Occiput-atlas-axis global manipulation
Other: Manual Therapy — All patients were assessed in the same conditions before the treatment, after the treatment (at 4 weeks), and at follow-up (after 8 weeks). Four treatment sessions (one session per week). Prior to each treatment session, the physiotherapist performed the vertebral artery test bilaterally, followed by a two-minute neck massage without lubricants and with no proven therapeutic effect, as a placebo for all study groups.
  The combination of both treatments aims to determine whether this combination has greater effects than the separate application of each treatment. After receiving the treatment, the subjects in the experimental groups stayed for five minutes in the supine resting position, in neutral ranges of cervical flexion, extension, lateral flexion and rotation.
  Arms: The combination of both treatments
Other: Placebo control — All patients were assessed in the same conditions before the treatment, after the treatment (at 4 weeks), and at follow-up (after 8 weeks). Four treatment sessions (one session per week). Prior to each treatment session, the physiotherapist performed the vertebral artery test bilaterally, followed by a two-minute neck massage without lubricants and with no proven therapeutic effect, as a placebo for all study groups.
  The control group received four sessions of placebo treatment, followed by ten minutes of resting position.
  Arms: control group

SUMMARY:
Background. Headache is one of the most common causes of consultation in primary health care and neurology in Europe. Cervical muscle tension can maintain a restriction of joint motion at the suboccipital level, facilitating the referred head pain.

Objective. To evaluate the effectiveness of two manual therapy treatments for tension-type headache.

Methods. A randomized double-blind clinical trial was conducted, for a period of 4 weeks and a follow-up at one month post-treatment. Eighty-four patients with tension-type headache were assigned to 4 groups (3 treatment groups and 1 control group). Treatments included manual therapy of suboccipital soft tissue inhibition, occiput-atlas-axis global manipulation, and a combination of both techniques. Outcome measures were: impact of headache, disability caused by headache, ranges of motion of the craniocervical junction, frequency and intensity of headache, and associated headache symptoms.

Results. After 8 weeks, there were significant improvements in impact of headache (p=0.01), disability (p=0.001), and craniocervical flexion (p=0.03) for the suboccipital soft tissue inhibition group; in headache impact and disability (p=0.000), pain intensity (p=0.02) and craniocervical flexion (p=0.004) and extension (p=0.04) for the occiput-atlas-axis group; and in impact (p=0.002), functional disability (p=0.000), headache frequency (p=0.002) and intensity (p=0.001), craniocervical flexion (p=0.008) and extension (p=0.003) and associated headache symptoms (p=0.01) for the combined therapy group, with effect sizes from medium to large.

Conclusions. Occiput-atlas-axis and combined therapy group treatments are more effective than suboccipital soft tissue inhibition for tension-type headache. The treatment with suboccipital soft tissue inhibition, despite producing less significant results, also has positive effects on different aspects of headache.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years, episodes of headaches lasting from 30 minutes to 7 days, headache having at least two of the following characteristics: *bilateral location

  * pressing non-pulsating quality
  * mild or moderate intensity
  * not aggravated by routine physical activity.
* Participants may present photophobia or phonophobia, nausea or vomiting, pericranial tenderness, with evolution of more than three months, and they must be under pharmacological control.

Exclusion Criteria:

* Patients with other types of headache
* Headache that is aggravated by head movements
* Metabolic disorders or musculoskeletal complaints previous neck trauma
* Vertigo
* Dizziness
* Arterial hypertension
* Advanced degenerative osteoarthritis
* Neck joint stiffness
* Signs of malignancy
* Pregnancy
* Patients with cardiac devices
* Patients in process of pharmacological adaptation, and excessive emotional tension

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2010-01; Primary Completion 2010-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Firstly, an individual clinical interview was conducted to collect socio-demographic data and characteristics of headache in a one-month base period (the previous 4 weeks) | up to 4 weeks
  This interview gathers information about age, sex, intensity and frequency of headache (with a Visual Analog Scale from 0 to 10), severity of pain (low, moderate, high), qualities of pain (Bilateral location of pain, Pulsating pressure, Not aggravated by physical activity, Photofobia/Phonofobia, Nausea/Vomiting, Pericranial tenderness), cranial location of pain, family history of headache, triggers, aggravating and pain-relieving factors, as well as any previous physiotherapy treatment for headache relief.

SECONDARY OUTCOMES:
Impact of headache on daily life(HIT-6) | up to 8 weeks
  It consists of 6 items each with 4 response options ranging from "never" (6 points) to "always" (13 points), and has shown high reliability in previous studies (alpha 0.87).
Headache Disability Inventory (HDI) | up to 8 weeks
  Two first items concerning the frequency and intensity of headaches and a questionnaire of 25 items assessing emotional and functional aspects with 4 possible response options, with an alpha reliability of 0.76-0.83
Headache pain intensity | up to 8 weeks
  rated daily by the patient on the 0-10 Visual Analogue Scale (VAS) (0 = no pain, 10 = most severe pain).
Ranges of motion of the craniocervical junction | up to 8 weeks
  measured with the CROM-device. This instrument has demonstrated a good intra-tester reliability for the movements of cervical flexion, extension, lateral flexion and rotation (ICC > 0.80) (ICC>0.80). However, not having found any previous studies about its reliability for the craniocervical junction (upper cervical joint), we performed -before using this device in our study- an inter-tester reliability analysis with our two examiners and 10 patients not participating in this study, which showed a Pearson's correlation of 0.98
Headache diary | up to 8 weeks
  During the four-week treatment period and in the follow-up phase, patients recorded on a daily basis the characteristics of headache with data regarding headache frequency and intensity, associated headache symptoms of photophobia or phonophobia, nausea or vomiting, and pericranial tenderness, completing a total of 7 weekly records.

CONTACTS AND LOCATIONS:
Overall Officials: Gemma Victoria Espí López, PhD, Principal Investigator — Physiotherapy Department. University of Valencia. Spain
Locations (1):
- Gemma V Espí López, Valencia, Valencia, Spain

REFERENCES:
- [Background] Castien RF, van der Windt DA, Grooten A, Dekker J. Effectiveness of manual therapy for chronic tension-type headache: a pragmatic, randomised, clinical trial. Cephalalgia. 2011 Jan;31(2):133-43. doi: 10.1177/0333102410377362. Epub 2010 Jul 20. PMID 20647241
- [Derived] Espi-Lopez GV, Gomez-Conesa A, Gomez AA, Martinez JB, Pascual-Vaca AO, Blanco CR. Treatment of tension-type headache with articulatory and suboccipital soft tissue therapy: A double-blind, randomized, placebo-controlled clinical trial. J Bodyw Mov Ther. 2014 Oct;18(4):576-85. doi: 10.1016/j.jbmt.2014.01.001. Epub 2014 Jan 10. PMID 25440210